CLINICAL TRIAL: NCT05922670
Title: The BH-Works Suicide Prevention Program for Sexual and Gender Minority Youth
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Collaborators: Drexel University (Other); Mazzoni Health Center (Unknown); Thomas Jefferson University (Other); Carilion Clinic (Other); Diversity Camp, Inc. (Unknown)
Responsible Party: Principal Investigator, Jody Russon, Assistant Professor, Virginia Polytechnic Institute and State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 22-079
Record Dates: First submitted 2023-05-16; First posted 2023-06-28 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Suicide; Engagement, Patient
Keywords: Sexual and Gender Minority Youth; Suicide Prevention Program; Effectiveness-Implementation Hybrid
MeSH Terms: conditions — Suicide; Patient Participation; Coitus | interventions — Sex

STUDY DESIGN:
Intervention Model Description: Behavioral health-Works (BH-Works) is a systems-level, multicomponent suicide prevention program designed for youth populations. The program includes two primary components, comprehensive web-based behavioral health screening (BHS), and an electronic referral system. This project will adapt and import this program into lesbian, gay, bisexual, transgender, and queer (LGBTQ) organizations. This project builds upon robust partnerships with two diverse LGBTQ organizations in Philadelphia, Pennsylvania and in rural Roanoke, Virginia and their behavioral health partners.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SGM BH-Works Implementation (Experimental): For this phase of the study, the adapted version of the BH-works program (SGM BH-Works) will be implemented into LGBTQ+ Community Organizations. The BH-Works program offers screening, training, and referral coordination.
  Interventions: Behavioral: The Behavioral Health-Works Suicide Prevention Program for Sexual and Gender Minority Youth

INTERVENTIONS:
Behavioral: The Behavioral Health-Works Suicide Prevention Program for Sexual and Gender Minority Youth — BH-Works is a web-based, comprehensive program for suicide prevention. The BH-Works program is a systems-level intervention that provides tools and resources to make organization adoption more feasible.
  Other Names: SGM BH-Works

SUMMARY:
Youth suicide is a serious public health concern. Compared to their heterosexual and cisgender peers, sexual and gender minority (SGM) adolescents report higher rates of suicidal ideation and suicide attempts. Unfortunately, many barriers complicate the implementation of suicide prevention in SGM communities. SGM youth often report feeling unwelcome in traditional behavioral health service organizations. Consequently, treatment attendance and retention remain low. Instead, this population generally seeks mental health services in community organizations for lesbian, gay, bisexual, transgender, and queer (LGBTQ) youth. These organizations are often unprepared for this clinical challenge. The Behavioral Health-Works (BH-Works) suicide risk management system may offer a potential solution to this problem. BH-Works is an evidence-based, comprehensive youth suicide prevention program. It offers support for policy development, staff training, suicide and behavioral health screening, technology-assisted safety planning, an electronic patient referral system, real-time data analytics for program monitoring, and a learning collaborative structure to support sustainability. All functions are supported on a web-based software platform that facilitates cross-system communication, implementation, adoption, and expansion. In this project, the investigators will adapt this program for LGBTQ organizations and test feasibility, acceptability and preliminary effectiveness. This project builds upon robust partnerships with two diverse LGBTQ organizations in Philadelphia, Pennsylvania and rural Southwest, Virginia) and their respective behavioral health (BH) partnering sites. To facilitate BH-Works adaptation for SGM adolescents, the investigators will employ the Enhancing Engagement trajectory from Lau's cultural adaptation framework. To pilot the program within LGBTQ organizations and their partners, the investigators will use an Effectiveness-Implementation Hybrid Type 2 design with a historical comparison group. Informed by the Consolidated Framework for Implementation Research, the investigators will also pilot test a sequenced implementation strategy. This strategy focuses on promoting engagement, building partnerships, and creating sustainability. In Years 1 and 2, the investigators will collect treatment as usual data, and work with their partners to adapt BH-Works policy, content, practices, and workflow. The investigators will also train staff/providers in suicide risk management, family engagement and affirmative care. In Years 3 and 4, the investigators will test the adapted SGM BH-Works Program and examine several essential program targets (training impact, partnership development, software usability) and outcomes (successful referral, program satisfaction, caregiver involvement, suicide identification).

DETAILED DESCRIPTION:
Suicide is the second leading cause of death for 15-to-24-year-olds in the United States (U.S.). Yet, only 14% of youth with suicidal ideation and 22% of those who make a suicide attempt, report receiving mental health services. The circumstances that sexual and gender minority (SGM) youth face are particularly alarming. Compared to their heterosexual and cisgender peers, SGM adolescents report far higher rates of suicidal ideation and suicide attempts. Consequently, adoption of effective suicide prevention programs, that increase identification and referral in organizations serving this population, are sorely needed.

Unfortunately, many barriers complicate the implementation of suicide prevention for SGM communities. SGM youth often report feeling unwelcome and misunderstood in traditional behavioral health service organizations. Consequently, treatment attendance and retention remain low. Instead, this population generally seeks mental health services in community organizations for lesbian, gay, bisexual, transgender, and queer (LGBTQ) youth. Unfortunately, these organizations are often unprepared for this clinical challenge. Specifically, they lack a) training in risk assessment, b) standardized screening tools, and c) access to behavioral health (BH) services that staff trust. In addition, staff in LGBTQ organizations express concern that many BH providers lack the SGM-sensitivity needed to work with this high risk, vulnerable population. Given these challenges, suicide prevention for SGM youth requires a multi-faceted program aimed to improve resources within these organizations and relationships between service systems.

A potential solution to this challenge is the Behavioral Health-Works (BH-Works) suicide risk management system. Similar to the identify, treat and refer structure of screening, brief intervention, and referral to treatment (SBIRT) for substance use, BH-Works includes support for policy development, staff training, suicide and behavioral health screening, technology-assisted safety planning, an electronic patient referral system, real-time data management for program monitoring, and a learning collaborative structure to support sustainability. All functions are supported on a web-based platform that facilitates cross-system communication, implementation, adoption, and expansion. BH-Works has been used in both clinical and non-clinical settings. In this project, the investigators will adapt BH-Works for SGM adolescents presenting in LGBTQ organizations and use data from the web-based screening and EMR systems to measure targets and outcomes. The investigators will employ the Enhancing Engagement trajectory, from Lau's cultural adaptation framework for this purpose. Lau recommends that adaptation of evidence-based treatments (EBTs) is necessary when contextual processes (e.g. discrimination, caregiver support, mistrust of health systems) contribute to unique vulnerabilities in specific populations, particularly those living in contexts where fewer specialized services exist. This project builds upon partnerships with two LGBTQ organizations in Philadelphia, and rural Southwest, Virginia) and their respective behavioral health (BH) partners.

The investigators will use an Effectiveness-Implementation Hybrid Type 2 design, with a historical comparison group, to test the feasibility, acceptability, and preliminary effectiveness of BH-Works within the LGBTQ organizations and their BH partners. Informed by the Consolidated Framework for Implementation Research (CFIR), the investigators will pilot test a sequenced implementation strategy. This strategy focuses on building partnerships and involves a) promoting engagement, b) strengthening relationships, and c) creating sustainability. In Year 1, the investigators will collect treatment as usual data, and work with stakeholders to adapt BH-Works policy, content, practices, and workflow. The investigators will also train staff in suicide risk management, family engagement, and affirmative care. In Years 2 and 3, the investigators will test the adapted SGM BH-Works Program and examine several essential program targets and outcomes, which are outlined in the aims.

Three aims focus on engagement, adaptation, and feasibility/acceptability of SGM BH-Works. Aim #1: Engage LGBTQ organization staff and partnering behavioral health providers. This aim focuses on: a) engaging a stakeholder advisory group, and b) initiating the implementation strategy. Aim #2: Adapt and pilot the BH-Works Program for LGBTQ organizations and partnering behavioral health sites. The adapted BH-Works Program will be implemented into LGBTQ organizations' workflow for a one-month open trial. Qualitative and quantitative data will be collected to evaluate initial feasibility and acceptability as well as to explore barriers and facilitators to usability in urban and rural organizations. The manual will undergo revisions. Aim #3: Test the feasibility, acceptability, and preliminary effectiveness of the SGM BH-Works Program compared to a historical control group. This quasi-experimental design will test the relationships between targets (training impact, partnership development, software usability) and outcomes (successful referral, program satisfaction, caregiver involvement, suicide identification). The proposed research responds to the growing national need to identify and refer vulnerable youth at risk for suicide.

Timeline: Control group data will be collected from month 5-18, while the investigators do manual and program adaptation (Aim #1). In months 19-24, the investigators will conduct the Zero Suicide evaluation, conduct trainings with LGBTQ organizations and BH site staff, pilot the program for a month, and gather initial feedback (focus groups) on the program to make final adaptations to the manual. Training consultations with staff will proceed bi-monthly through month 41 (Aim #2). In months 25-41, the investigators will run the program and collect satisfaction (consumers), feasibility, acceptability, and preliminary effectiveness data (Aim #3). In months 42-44, the investigators will do closing focus groups with staff, administrators, caregivers, and patients at all sites. Following this, the investigators will write up manuscripts and an R01 to test the SGM BH-Works program on a larger scale. Research aims for this three-year project will be completed with the addition of a fourth no cost extension year.

Procedure: Procedures are broken down by aim.

Aim #1: Engage LGBTQ organization staff and partnering behavioral health providers. This aim focuses on: a) engaging a stakeholder advisory group, and b) initiating the implementation strategy.

Administrative stakeholder participants have already agreed to participate in this research and serve as Co-Is on the project. LGBTQ staff/behavioral health provider participants will be recruited by leadership to participate in this project. The investigators expect to include 4-8 staff/providers/administrators at each site. Consenting processes will occur immediately before initial evaluation activities and the first trainings begins. Each agency reports having at least 4 to 6 intake workers and all will be trained in the program. These staff members will complete assessments at the beginning of the study and then five times over the course of years 2-4. They will participate in a final interview after the one month pilot period and at the end of the study.

Engage advisory board and workgroup. A local and national advisory board will serve as project collaborators. This group includes academics, educators, administrators, practicing professionals, and community members who are committed to SGM health (see letters of support and commitment). The principal investigator's partners at will assist in identifying SGM youth and their caregivers to serve on the board. The investigators' collaboration with an organizing body for LGBTQ community centers in the world, will have a central role in steering this project. A smaller workgroup will consist of project investigators, leadership from partnering sites, and an implementation consultant. The advisory board meets every two-three months throughout the project.

Aim #2: Adapt and pilot the BH-Works Program for LGBTQ organizations and partnering behavioral health sites. The adapted BH-Works Program will be implemented into LGBTQ organizations' workflow for a one-month open trial. Qualitative and quantitative data will be collected to evaluate initial feasibility and acceptability as well as to explore barriers and facilitators to usability in urban and rural organizations. The manual will undergo revisions.

Adaptation process. The investigators will employ Lau's framework for the cultural adaptations of evidence-based treatments (EBTs). Lau recommends that adaptation of EBTs is necessary when contextual processes (e.g. discrimination, caregiver support, mistrust of health systems) contribute to unique vulnerabilities in specific populations, such as SGM youth (particularly those living in rural contexts where fewer specialized LGBTQ services exist). In this project, the investigators focus on Lau's Enhancing Engagement trajectory of adaptation work. As such, the workgroup will focus on generating BH-Works program adaptations that will increase social validity, a potential target for increasing engagement. The role of the workgroup is essential in the adaptation process. The investigators expect this group will increase the social validity of the program by helping us adapt the screening language to be more affirmative, better manage matters of pronoun use, and address concerns about discrimination in standard operating procedures.

Adolescent, emerging adult, and caregiver participation in the pilot process mirrors what is described below in Aim #3. Following the Aim #2 pilot of the BH-Works program, organization staff, patients and caregivers will be invited to participate in a focus group to discuss features of the BH-Works program that they find appealing and unappealing, as well as suggestions for improvement. Responses will be consolidated across group and location type (urban vs. rural).

Aim #3: Test the feasibility, acceptability, and preliminary effectiveness of the SGM BH-Works Program compared to a historical control group. This quasi-experimental design will test the relationships between targets (training impact, partnership development, software usability) and outcomes (successful referral, program satisfaction, caregiver involvement, suicide identification). The proposed research responds to the growing national need to identify and refer vulnerable youth at risk for suicide.

Treatment as usual data will be extracted as de-identified medical records data at the LGBTQ organizations. Data will be collected on the number of patients who were a) assessed for suicide, b) identified as at risk for suicide, and c) referred for behavioral health services. As part of standard care procedures, staff currently conduct a one week follow up call on any patient referred for services, asking if they attended and about their experience. To facilitate comparison with the intervention group, the investigators will ask LGTBQ staff members to include 4-item Acceptability of Intervention Measure on their experience with a) the referral process, and b) their first behavioral health appointment (see measures section).

Treatment as usual data for the control group will be extracted as de-identified records data at the LGBTQ organizations in Years 1 and 2. Data will be collected on the number of patients who were a) assessed for suicide, b) identified as at risk for suicide, and c) referred for behavioral health services. To facilitate comparison with the intervention group, the investigators will ask LGTBQ staff members to include 4-item Acceptability of Intervention Measure (AIM) on their experience with a) the referral process, and b) their first behavioral health appointment.

Once the BH-Works program is implemented in Years 2 and 3, adolescent consent will begin at the point of screening. The BH-Works screening tool will be included in the standard of care procedures. However, the principal investigator's Institution Review Board (IRB) has approved a brief consent at the beginning of the screen asking permission to use de-identified screening data for research; 90% of patients agree to participate. At the end of the BHS, participants complete a brief satisfaction measure about their experience with the screening tool. This is included as part of the screening process for ongoing quality improvement (QI) purposes. In investigators' past studies, if patients endorse any level of current suicidal ideation, a consent form is automatically presented at the end of the screening asking permission to follow up with the adolescent in one week and one month to see if services were recommended and obtained. However, in this study, the LGBTQ agencies already do a standard of care follow up call to see if patients went to services. As such, they will ask if the research team can call to follow up with them about participating in an interview about seeking services. Consent for participation in this follow-up assessment will occur in the first part of the meeting. In both PA and VA, youth, ages 14 and older, can seek their own mental health services without parental consent. At partnering LGBTQ organizations, many adolescents do not want their parents involved. These youth can still participate in this project without involving their parent, even though caregiver engagement will be encouraged.

Caregivers will be recruited in a similar fashion as adolescent patients. After receiving family engagement training, it is expected that staff will be able to engage approximately 50-60% patients' caregivers in the referral process. If caregivers have been engaged, staff will ask if the research team can contact them about participating in a follow up research assessment about seeking help. As with patient participants, caregivers will be contacted to set up a 60-minute meeting a week after their child was screened and referred. Caregivers will provide consent at the beginning of the meeting. The investigators will not exclude caregivers from participation if their adolescent chooses not to participate (and vice versa). It is likely these individual participants can offer important perspectives on screening and referral processes.

ELIGIBILITY:
Inclusion Criteria:

1. youth must be seeking services at the participating LGBTQ organizations.
2. youth must endorse current suicidal ideation on the BHS.

Exclusion Criteria:

1. youth lack enough English-language proficiency to complete the BH-Works program
2. youth are not capable of understanding the requirements for study participation

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 260 (Estimated)
Dates: Start 2022-08-24 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-24 (Estimated)

PRIMARY OUTCOMES:
Successful Referral (Youth attends a first behavioral health session with a behavioral health provider at the recommendation of LGBTQ organization staff) | Self and staff report (medical records) collected within one week to one month after participant enrolls in study and completes the behavioral health screen.
  Youth and staff report (medical records) indicate that the youth has attended a first behavioral health appointment at the behavioral health site that LGBTQ organization staff referred them to. This data will be recorded dichotomously (no= 0; yes=1).
Acceptability of Intervention Measure (AIM) | Self report collected within one week to one month after participant enrolls in study and completes the behavioral health screen.
  Using this 4-item measure, youth will report on their perceptions of the acceptability (satisfaction) for the screening and referral process occurring with LGBTQ community staff as well as for their first appointment with the behavioral health provider to whom they were referred. The Acceptability of Intervention Measure is scored on a 5-point Likert scale (1 = strongly disagree, 5 = strongly agree), then either averaged [total score 1-5] or reported as a total [total score 4-20].
Caregiver Involvement (Caregiver was observed by LGBTQ organization staff as being involved in the screening and referral process with their youth) | Staff report collected within one week to one month after participant enrolls in study and completes the behavioral health screen.
  LGBTQ organization staff will indicate whether a caregiver has been involved in the screening and referral process taking place at LGBTQ organizations. This data will be recorded dichotomously (no= 0; yes=1).
Behavioral Health Screen Suicide Subscale | Collected at time of study enrollment.
  The suicide subscale of the behavioral health screen consists of four items asking youth about suicide ideation and behavior. Item responses followed a three-point scale: no reported symptoms, moderate symptoms, or severe symptoms. Higher scores indicate higher risk for suicide.

SECONDARY OUTCOMES:
Gatekeeper Behavior Scale (Adapted Version) | Completed pre- and post- training during year 2, and every 6 months during the 18-month experimental phase.
  The investigator's adapted version of the GBS consists of subscales (knowledge, attitudes, preparedness, liklihood, self-efficacy).This adapted measure has demonstrated strong psychometrics. The measure is scored by standardizing the mean score of the subscales. Total scores range between 0 and 100, with a higher score indicating greater liklihood of 'engaging in gatekeeper intervention behaviors.' For this proposed study, the investigators will also adapt this scale to measure the impact the affirmative care training curriculum.
Partnership Development Items | Completed pre- and post- training during year 2, and every 6 months during the 18-month experimental phase.
  Partnership development will be measured by a brief questionnaire (to be developed in collaboration with our advisory board). For LGBTQ staff, the investigators will ask questions about partnerships with behavioral health partners (e.g., to what extent do you feel confident behavioral health partners can work with LGBTQ youth?). Questions will be measured as single items with higher scores indicating stronger partnerships.
Software Usability Survey | Completed pre- and post- training during year 2, and every 6 months during the 18-month experimental phase.
  The Software Usability Measurement Interview will be used to measure usability for staff/providers. It has 50 Likert-scale items and takes about 5 minutes. It addresses a standard set of usability factors consisting of: Affect, Control, Helpfulness, Learnability, and Efficiency. The quantitative goal is for each factor to achieve a score of at least 80% of the maximum possible score. Progress over the course of the pilot period meeting these goals will be tracked by the successive usability scores.
  The SUMI consists of 50 attitude statements, to each of which the user may respond 'agree', 'don't know', or 'disagree'. SUMI is scored and interpreted with reference to a standardization database representing a mixed bag of software products (ranging from CAD to office products). This database is updated yearly. The global usability score is set to an average score of 50 with scores above 50 indicating more user-friendly and below as less user-friendly.

CONTACTS AND LOCATIONS:
Overall Officials: Jody M. Russon, PhD, Principal Investigator — Virginia Polytechnic Institute and State University
Locations (5):
- United States (5):
  - Drexel University, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Mazzoni Center, Philadelphia, Pennsylvania
  - Carilion Clinic, Roanoke, Virginia
  - Diversity Camp, Inc., Roanoke, Virginia

IPD SHARING:
Plan to Share IPD: Yes
All youth participants will agree to the sharing of data results with the (National Institute of Mental Health (NIMH) Data Archive (NDA). All data will be de-identified prior to receipt by the repository, but the information needed to generate a (global unique identifier) GUID will be collected for each participant. The proposed research will also involve collecting data from approximately 50-60% of caregivers whose adolescents participate in the research. Demographic information from these participating caregivers will be shared using the procedures described for adolescent participants above.
Time Frame: If funded, within 6 months of the Notice of Award date the investigators will submit a Data Submission Agreement signed by the principal investigator and an institutional business official, as well as define and complete the Data Expected section of this project. Uploads of all initial demographic and clinical data will be completed by the next submission cycle deadline following the initiation of data collection of clinical assessments outlined in the timeline for this project. Clinical data collection, therefore, will occur when the pilot phase begins, month 11 (July 2023) of the project. The next submission cycle deadline following July 2023 would be January 15th, 2024. Subsequent data uploads will be harmonized, validated, and submitted biannually on the standard January 15th and July 15th submission deadlines.

REFERENCES:
- [Background] Hoyert DL, Xu J. Deaths: preliminary data for 2011. Natl Vital Stat Rep. 2012 Oct 10;61(6):1-51. PMID 24984457
- [Background] Lau AS. Making the case for selective and directed cultural adaptations of evidence-based treatments: Examples from parent training. Clinical psychology: Science and practice. 2006;13(4):295.
- [Background] Curran GM, Bauer M, Mittman B, Pyne JM, Stetler C. Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. Med Care. 2012 Mar;50(3):217-26. doi: 10.1097/MLR.0b013e3182408812. PMID 22310560
- [Background] Nock MK, Green JG, Hwang I, McLaughlin KA, Sampson NA, Zaslavsky AM, Kessler RC. Prevalence, correlates, and treatment of lifetime suicidal behavior among adolescents: results from the National Comorbidity Survey Replication Adolescent Supplement. JAMA Psychiatry. 2013 Mar;70(3):300-10. doi: 10.1001/2013.jamapsychiatry.55. PMID 23303463
- [Background] Bauer GR, Scheim AI, Pyne J, Travers R, Hammond R. Intervenable factors associated with suicide risk in transgender persons: a respondent driven sampling study in Ontario, Canada. BMC Public Health. 2015 Jun 2;15:525. doi: 10.1186/s12889-015-1867-2. PMID 26032733
- [Background] Haas AP, Eliason M, Mays VM, Mathy RM, Cochran SD, D'Augelli AR, Silverman MM, Fisher PW, Hughes T, Rosario M, Russell ST, Malley E, Reed J, Litts DA, Haller E, Sell RL, Remafedi G, Bradford J, Beautrais AL, Brown GK, Diamond GM, Friedman MS, Garofalo R, Turner MS, Hollibaugh A, Clayton PJ. Suicide and suicide risk in lesbian, gay, bisexual, and transgender populations: review and recommendations. J Homosex. 2011;58(1):10-51. doi: 10.1080/00918369.2011.534038. PMID 21213174
- [Background] Perez-Brumer A, Day JK, Russell ST, Hatzenbuehler ML. Prevalence and Correlates of Suicidal Ideation Among Transgender Youth in California: Findings From a Representative, Population-Based Sample of High School Students. J Am Acad Child Adolesc Psychiatry. 2017 Sep;56(9):739-746. doi: 10.1016/j.jaac.2017.06.010. Epub 2017 Jul 5. PMID 28838578
- [Background] Toomey RB, Syvertsen AK, Shramko M. Transgender Adolescent Suicide Behavior. Pediatrics. 2018 Oct;142(4):e20174218. doi: 10.1542/peds.2017-4218. Epub 2018 Sep 11. PMID 30206149
- [Background] Guss CE, Woolverton GA, Borus J, Austin SB, Reisner SL, Katz-Wise SL. Transgender Adolescents' Experiences in Primary Care: A Qualitative Study. J Adolesc Health. 2019 Sep;65(3):344-349. doi: 10.1016/j.jadohealth.2019.03.009. Epub 2019 Jun 18. PMID 31227384
- [Background] Qureshi RI, Zha P, Kim S, Hindin P, Naqvi Z, Holly C, Dubbs W, Ritch W. Health Care Needs and Care Utilization Among Lesbian, Gay, Bisexual, and Transgender Populations in New Jersey. J Homosex. 2018;65(2):167-180. doi: 10.1080/00918369.2017.1311555. Epub 2017 May 8. PMID 28481718
- [Background] Olson-Kennedy J, Cohen-Kettenis PT, Kreukels BP, Meyer-Bahlburg HF, Garofalo R, Meyer W, Rosenthal SM. Research priorities for gender nonconforming/transgender youth: gender identity development and biopsychosocial outcomes. Curr Opin Endocrinol Diabetes Obes. 2016 Apr;23(2):172-9. doi: 10.1097/MED.0000000000000236. PMID 26825472
- [Background] Fish JN, Moody RL, Grossman AH, Russell ST. LGBTQ Youth-Serving Community-Based Organizations: Who Participates and What Difference Does it Make? J Youth Adolesc. 2019 Dec;48(12):2418-2431. doi: 10.1007/s10964-019-01129-5. Epub 2019 Oct 12. PMID 31606828
- [Background] Pachankis JE, Clark KA, Jackson SD, Pereira K, Levine D. Current Capacity and Future Implementation of Mental Health Services in U.S. LGBTQ Community Centers. Psychiatr Serv. 2021 Jun;72(6):669-676. doi: 10.1176/appi.ps.202000575. Epub 2021 Apr 22. PMID 33882684
- [Background] Allen KD, Hammack PL, Himes HL. Analysis of GLBTQ youth community-based programs in the United States. J Homosex. 2012;59(9):1289-306. doi: 10.1080/00918369.2012.720529. PMID 23101498
- [Background] Skaer TL, Sclar DA, Robison LM. Trends in prescriptions for antidepressant pharmacotherapy among US children and adolescents diagnosed with depression, 1990 through 2001: an assessment of accordance with treatment recommendations from the American Academy of Child and Adolescent Psychiatry. Clin Ther. 2009 Jun;31 Pt 1:1478-87. doi: 10.1016/j.clinthera.2009.07.002. PMID 19698905
- [Background] Wintersteen MB, Diamond GS. Youth suicide prevention in primary care: A model program and its impact on psychiatric emergency referrals. Clinical Practice in Pediatric Psychology. 2013 Sep;1(3):295.
- [Background] Williams SB, O'Connor EA, Eder M, Whitlock EP. Screening for child and adolescent depression in primary care settings: a systematic evidence review for the US Preventive Services Task Force. Pediatrics. 2009 Apr;123(4):e716-35. doi: 10.1542/peds.2008-2415. PMID 19336361
- [Background] Fein JA, Pailler ME, Barg FK, Wintersteen MB, Hayes K, Tien AY, Diamond GS. Feasibility and effects of a Web-based adolescent psychiatric assessment administered by clinical staff in the pediatric emergency department. Arch Pediatr Adolesc Med. 2010 Dec;164(12):1112-7. doi: 10.1001/archpediatrics.2010.213. PMID 21135339
- [Background] Diamond G, Levy S, Bevans KB, Fein JA, Wintersteen MB, Tien A, Creed T. Development, validation, and utility of internet-based, behavioral health screen for adolescents. Pediatrics. 2010 Jul;126(1):e163-70. doi: 10.1542/peds.2009-3272. Epub 2010 Jun 21. PMID 20566613
- [Background] Diamond GS, Herres JL, Krauthamer Ewing ES, Atte TO, Scott SW, Wintersteen MB, Gallop RJ. Comprehensive Screening for Suicide Risk in Primary Care. Am J Prev Med. 2017 Jul;53(1):48-54. doi: 10.1016/j.amepre.2017.02.020. Epub 2017 Apr 11. PMID 28410860
- [Background] Substance Abuse and Mental Health Services Administration. (2012). Screening, Brief Intervention, and Referral to Treatment (SBIRT). U.S. Department of Health and Human Services. https://www.samhsa.gov/sbirt
- [Background] Damschroder LJ, Aron DC, Keith RE, Kirsh SR, Alexander JA, Lowery JC. Fostering implementation of health services research findings into practice: a consolidated framework for advancing implementation science. Implement Sci. 2009 Aug 7;4:50. doi: 10.1186/1748-5908-4-50. PMID 19664226
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- [Background] Braun V, Clarke V. Using thematic analysis in psychology. Qualitative research in psychology. 2006 Jan 1;3(2):77-101.
- [Background] Diamond GM, Shilo G, Jurgensen E, D'Augelli A, Samarova V, White K. How depressed and suicidal sexual minority adolescents understand the causes of their distress. Journal of Gay & Lesbian Mental Health. 2011 Mar 31;15(2):130-51.
- [Background] Diamond G, Kodish T, Ewing ESK, Hunt QA, Russon JM. Family processes: Risk, protective and treatment factors for youth at risk for suicide. Aggress Violent Behav. 2022 May-Jun;64:101586. doi: 10.1016/j.avb.2021.101586. Epub 2021 Mar 9. PMID 35662798
- [Background] Albright GL, Davidson J, Goldman R, Shockley KM, Timmons-Mitchell J. Development and Validation of the Gatekeeper Behavior Scale. Crisis. 2016 Jul;37(4):271-280. doi: 10.1027/0227-5910/a000382. Epub 2016 Jun 1. PMID 27245815
- [Background] Asarnow JR, Miranda J. Improving care for depression and suicide risk in adolescents: innovative strategies for bringing treatments to community settings. Annu Rev Clin Psychol. 2014;10:275-303. doi: 10.1146/annurev-clinpsy-032813-153742. Epub 2014 Jan 16. PMID 24437432
- [Background] Coleman N. SUMI (Software Usability Measurement Inventory) as a knowledge elicitation tool for improving usability. 1993; Unpublished BA Honours thesis, Dept. Applied Psychology, University College Cork, Ireland.
- [Background] Fish JN. Future Directions in Understanding and Addressing Mental Health among LGBTQ Youth. J Clin Child Adolesc Psychol. 2020 Nov-Dec;49(6):943-956. doi: 10.1080/15374416.2020.1815207. Epub 2020 Oct 19. PMID 33074740
- [Background] Guo W, Ratcliffe SJ, Have TT. A random pattern-mixture model for longitudinal data with dropouts. Journal of the American Statistical Association. 2004 Dec 1;99(468):929-37.
- [Background] Hedeker D, Gibbons RD. Application of random-effects pattern-mixture models for missing data in longitudinal studies. Psychological methods. 1997 Mar;2(1):64.
- [Background] Kano M, Silva-Banuelos AR, Sturm R, Willging CE. Stakeholders' Recommendations to Improve Patient-centered "LGBTQ" Primary Care in Rural and Multicultural Practices. J Am Board Fam Med. 2016 Jan-Feb;29(1):156-60. doi: 10.3122/jabfm.2016.01.150205. PMID 26769889
- [Background] Raudenbush SW, Bryk AS. Hierarchical linear models: Applications and data analysis methods. sage; 2002.
- [Background] Richards JE, Simon GE, Boggs JM, Beidas R, Yarborough BJH, Coleman KJ, Sterling SA, Beck A, Flores JP, Bruschke C, Grumet JG, Stewart CC, Schoenbaum M, Westphal J, Ahmedani BK. An implementation evaluation of "Zero Suicide" using normalization process theory to support high-quality care for patients at risk of suicide. Implement Res Pract. 2021 Jan 1;2:26334895211011769. doi: 10.1177/26334895211011769. Epub 2021 May 24. PMID 34447940
- [Background] Russon J, Smithee L, Simpson S, Levy S, Diamond G. Demonstrating Attachment-Based Family Therapy for Transgender and Gender Diverse Youth with Suicidal Thoughts and Behavior: A Case Study. Fam Process. 2022 Mar;61(1):230-245. doi: 10.1111/famp.12677. Epub 2021 May 27. PMID 34046893
- [Background] Taliaferro LA, Muehlenkamp JJ. Nonsuicidal Self-Injury and Suicidality Among Sexual Minority Youth: Risk Factors and Protective Connectedness Factors. Acad Pediatr. 2017 Sep-Oct;17(7):715-722. doi: 10.1016/j.acap.2016.11.002. PMID 28865597
- [Background] Wallerstein N, Duran B. Community-based participatory research contributions to intervention research: the intersection of science and practice to improve health equity. Am J Public Health. 2010 Apr 1;100 Suppl 1(Suppl 1):S40-6. doi: 10.2105/AJPH.2009.184036. Epub 2010 Feb 10. PMID 20147663